CLINICAL TRIAL: NCT03549754
Title: Real-world Multinational Registry to Determine Management and Quality of Care of Patients With Type 2 Diabetes, Hypertension, Heart Failure and/or Chronic Kidney Diseases
Brief Title: iCaReMe Global Registry
Acronym: iCaReMe
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00044
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Hypertension; Chronic Kidney Disease; Heart Failure
Keywords: Registry; Type 2 Diabetes; T2DM; Chronic Kidney Disease; CKD; Hypertension; HTN; Adult population; Heart Failure; HF; Early cardiorenal complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Renal Insufficiency, Chronic; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To provide real world data on patient characteristics, disease management, healthcare utilization, and outcomes in patients with type 2 diabetes, Hypertension, Heart failure and/or Chronic kidney diseases

DETAILED DESCRIPTION:
The registry intends to provide real world data on patient management and quality of care for patients with T2DM, hypertension, heat failure and chronic kidney disease in clinical practice in many countries. To bridge this gap an observational voluntary registry is set up to capture real world data on patient characteristics, disease management, healthcare utilization, and outcomes in patients with type 2 diabetes, Hypertension, Heart Failure and Chronic Kidney Disease. Multinational, observational registry utilizing a cloud-based eCRF, for prospective and retrospective data collection, accessible to investigators and Scientific Committee. This registry will be open to all physicians managing T2DM, HTN, HF or CKD across the world

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years or older
2. Having type 2 diabetes, Hypertension, Heart Failure and/or chronic kidney disease
3. Providing written informed consent to participate in the registry

Exclusion Criteria:

1. Having a life-threatening co-morbidity with life expectancy below 1 year
2. Participating in an interventional trial requiring informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with type 2 diabetes, Hypertension, Heart Failure and/or chronic kidney disease
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2018-02-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Provide real world data on patient characteristics | Average of 3 years through study completion
  Disease control (e.g. achievement of glycated hemoglobin target and incidence of hypoglycemic events) Management of micro- and/or macrovascular complications Management of associated risk factors (e.g. hypercholesterolemia and hypertension) Current diabetes, CKD and HF treatments Concomitant medications
2. Provide real world data on disease management | Average of 3 years through study completion
  Disease control (e.g. achievement of glycated hemoglobin target and incidence of hypoglycemic events) Management of micro- and/or macrovascular complications Management of associated risk factors (e.g. hypercholesterolemia and hypertension) Current diabetes treatments Concomitant medications
3. Provide real world data on healthcare utilization | Average of 3 years through study completion
  Number of diabetes, Chronic Kidney Disease(CKD) and Heart Failure(HF)-related visits to a physician not at study site Number of urgent care visits for diabetes Number of diabetes, CKD and HF-related hospital emergency department visits and reason(s) for visits Number of hospitalizations, lengths of stay, and reasons for hospitalizations
4. Provide real world data on quality of care indicators | Average of 3 years through study completion
  Smoking cessation Eye and foot examinations Dietary counselling
Provide real world data on cardiovascular outcomes in patients with type 2 diabetes; Chronic Kidney Disease and Heart Failure | Average of 3 years through study completion
  All-cause and cause-specific deaths and hospitalizations, including recurrent events
6. Provide real world data on renal outcomes and other microvascular complications in patients with type 2 diabetes and Heart Failure | Average of 3 years through study completion
  All-cause and cause-specific deaths and hospitalizations, including recurrent events

CONTACTS AND LOCATIONS:
Locations (47):
- Brazil (13):
  - Research Site, Fortaleza, Ceará
  - Research Site, Colatina, Espírito Santo (ES)
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Brasília, Federal District
  - Research Site, Poços de Caldas, Minas Gerais
  - Research Site, Campina Grande do Sul, Paraná
  - Research Site, Teresina, Piauí (PI)
  - Research Site, Santa Cruz do Sul, Rio Grande Do Sul (RS)
  - Research Site, Goiânia, State of Goiás
  - Research Site, Joinville, State of Santa Catarina
  - Research Site, Bragança Paulist, São Paulo
  - Research Site, São Caetano do Sul, São Paulo
  - Research Site, São Paulo
- Research Site, Providencia, Santiago Metropolitan, Chile
- Research Site, Abidjan, Côte d’Ivoire
- Research Site, Wan Chai District, Hong Kong
- Research Site, Ahmedabad, India
- Research Site, Sunkar, Iraq
- Research Site, Almaty, Kazakhstan
- Research Site, Nairobi, Kenya
- Malaysia (2):
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Lumpur, Selangor
- Mexico (5):
  - Research Site, León, Guanajuato
  - Research Site, Colonia Doctores Neighborhood
  - Research Site, Iztapalapa
  - Research Site, Mexico City
  - Research Site, México
- Nigeria (2):
  - Research Site, Gwagwalada
  - Research Site, Kano
- South Africa (3):
  - Research Site, Florida
  - Research Site, Parow
  - Research Site, Umhlanga
- Taiwan (7):
  - Research Site, Niaosong Dist, Kaohsiung
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan
- Ukraine (7):
  - Research Site, Dnipro, Dnipropetrovsk Oblast
  - Research Site, Kharkiv, Kharkivs’ka Oblast’
  - Research Site, Kyiv, Kyiv Oblast
  - Research Site, Vinnytsia, Vinnytsia Oblast
  - Research Site, Lutsk, Volyn Oblast
  - Research Site, Uzhhorod, Zakarpattia Oblast
  - Research Site, Zaporizhzhia, Zaporizhzhia Oblast
- Research Site, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home